CLINICAL TRIAL: NCT01143584
Title: Efficacy of Rapid Escalation of Cabergoline in Comparison to Conventional Dosing in Prolactin Secreting Macroadenomas.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Anil Bhansali, Postgraduate Institute of Medical Education and Research
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: prlcab2020
Record Dates: First submitted 2010-06-01; First posted 2010-06-14 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-05

CONDITIONS: Macroprolactinoma
Keywords: Prolactin; Cabergoline; Macroadenomas; escalation
MeSH Terms: conditions — Prolactinoma | interventions — Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapid escalation (Experimental): Weekly escalation of cabergoline dose in macroprolactinomas Start with 1 mg/week. increase by 1mg/wk every week till 4 weeks. after 4 weeks Cabergoline dose would be increased @1mg/wk every 4 weekly till normalization of prolactin and >50% decrease in tumor volume from baseline.
  Interventions: Drug: cabergoline
- Conventional escalation (Active Comparator): Conventional escalation of cabergoline
  In the Conventional escalation group schedule of cabergoline dosing will be 0.5 mg once a week for 4 weeks. Cabergoline will be incrementally dose adjusted on the basis of individual Prolactin values till amelioration of hyper prolactinemia @ 0.5 mg/wk every 4 weeks, till 24 weeks or till primary endpoint.
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Cabergoline — In the Conventional escalation group Cabergoline 0.5 mg once a week for 4 weeks and further will be incrementally dose adjusted on the basis of individual PRL values until amelioration of hyper prolactinemia @ 0.5 mg/wk every 4 weeks, till 24 weeks or until primary endpoint.
  Cabergoline will be maintained at the dose at which PRL will be first normalized till primary end point.
  Arms: Conventional escalation
Drug: cabergoline — In the Rapid escalation group schedule of cabergoline dosing will be as follows:
  Begin with 0.5 mg twice a week
  1. mg twice a week - second week 1.5 mg twice a week - third week
  2. mg twice a week - fourth week
  4mg/wk would be continued for next 4 weeks. If prolactin does not normalize by 8 weeks, a repeat hike in dose of 1mg/wk will be done every 4 weekly until normalization of prolactin levels and also >50% decrease in tumor volume. Ceiling dose of Cabergoline will be 12mg/wk.
  Other Names: cabergoline dopamine agonist
  Arms: Rapid escalation

SUMMARY:
To study the effects of rapid escalation of Cabergoline in comparison to conventional dosing in macroprolactinomas. Rapid escalation of cabergoline may help in earlier normalization of prolactin and shrinkage of tumor mass, and thus decrease the cumulative dose of cabergoline altogether.

DETAILED DESCRIPTION:
The efficacy of cabergoline is dose related and determined by percentage of Dopamine 2 receptor occupancy and prolonged receptor affinity. Activation of membrane receptors and target cell responses is proportional to the degree of receptor occupancy. Greater the drug concentration, greater is the binding and receptor occupancy and greater is the efficacy of the drug. Receptor occupancy can be increased either by using high dose of cabergoline or by rapid escalation of cabergoline. The patients, who respond to increasing dosages of cabergoline, probably do so by increased receptor occupancy with higher doses.

Rapid escalation of doses of cabergoline is another approach to increase the drug concentration and increase the occupancy of the receptor. Earlier decrease in serum prolactin levels with rapid escalation may help in reducing the cumulative dose of cabergoline and total duration of treatment. Though studies with high doses of cabergoline have been performed in prolactinomas with normalization of prolactin levels in almost 100%, but systematic studies using rapid escalation of cabergoline in prolactinomas are lacking except the one by Bhansali et al. In their study, serum prolactin became normal in 93 per cent of the patients with a mean duration of 8.2 wk. The mean decrease in serum prolactin was 99 per cent by four weeks, however a similar decrease (93 to 99%) in prolactin was achieved in other studies with a time lag of 48 to 160 wk. This supports the notion that rapid hike in doses of cabergoline decreases serum prolactin levels faster and it becomes normal in the majority of patients earlier6. However it was an uncontrolled study with limited number of subjects.

Therefore present study was planned to study the efficacy of rapid escalation of Cabergoline versus conventional dosing in patients with macroprolactinomas. Rapid escalation of cabergoline dose may help in earlier normalization of prolactin and shrinkage of tumor mass, and thus decrease the cumulative dose of cabergoline altogether.

ELIGIBILITY:
Inclusion Criteria:

Males or females presenting with

1. Prolactin secreting macroadenomas (≥10 mm maximum diameter)
2. With/without visual complaints
3. With /without parasellar or suprasellar extension
4. Treatment Naïve

Exclusion Criteria:

1. On treatment with dopamine agonists.
2. Taking other drugs influencing prolactin Levels.
3. Systemic disease like Chronic Kidney Disease, Chronic Lung Disease
4. Other secondary causes of hyperprolactinemia.
5. Prolactin secreting microadenomas
6. Pregnancy during follow up
7. Prolactinoma as part of MEN-1 Syndrome
8. History suggestive of recent apoplexy (3 months)
9. Contraindication to cabergoline therapy like pre existing psychosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Normoprolactinemia | 1 year
  Duration for normalization of serum prolactin and decrease in tumor volume >50 % from baseline.

SECONDARY OUTCOMES:
Duration for resolution of Hypogonadism | 1 year
  Duration for resolution of hypogonadism in males as defined by normal serum total testosterone 9.9-27.8nmol/L and aging male study score(AMS). In females duration to acheive regular menstrual cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Bhansali, MD DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh; Pinaki Dutta, MD DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Rama Walia, MD DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Paramjeet Singh, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Vishali Gupta, MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Rajesh Vijaiwergiya, MD DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Ashu Rastogi, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Naresh Sachdeva, PhD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Rastogi A, Bhansali A, Dutta P, Singh P, Vijaivergiya R, Gupta V, Sachdeva N, Bhadada SK, Walia R. A comparison between intensive and conventional cabergoline treatment of newly diagnosed patients with macroprolactinoma. Clin Endocrinol (Oxf). 2013 Sep;79(3):409-15. doi: 10.1111/cen.12149. Epub 2013 Jul 2. PMID 23347435